CLINICAL TRIAL: NCT07316660
Title: Palmitoylethanolamide Versus Ibuprofen for Acute Postoperative Pain After Extracorporeal Shock Wave Lithotripsy: A Randomized Trial
Brief Title: Palmitoylethanolamide vs Ibuprofen for Pain After ESWL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Samar Rafik Mohamed Amin, assistant professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC.19.10.2025
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Pain After Extracorporeal Shock Wave Lithotripsy; Palmitoylethanolamide
MeSH Terms: interventions — palmidrol; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palmitoylethanolamide Group (Experimental): Participants assigned to this arm will receive oral palmitoylethanolamide for management of acute postoperative pain following extracorporeal shock wave lithotripsy (ESWL). Rescue analgesia will be available if required.
  Interventions: Drug: Palmitoylethanolamide (PEA)
- Ibuprofen Group (Active Comparator): Participants assigned to this arm will receive oral ibuprofen for management of acute postoperative pain following extracorporeal shock wave lithotripsy (ESWL). Rescue analgesia will be available if required.
  Interventions: Drug: Ibuprofen (Brufen®)

INTERVENTIONS:
Drug: Palmitoylethanolamide (PEA) — Palmitoylethanolamide (PEA) will be administered orally at a dose of 600 mg approximately 60 minutes before ESWL, followed by 600 mg every 8 hours for the first 24 hours after the procedure (total of three doses). PEA will be provided as a micronized or ultramicronized formulation. Participants will be allowed to receive rescue analgesia according to the study protocol if pain is not adequately controlled.
  Arms: Palmitoylethanolamide Group
Drug: Ibuprofen (Brufen®) — Ibuprofen will be administered orally at a dose of 400 mg approximately 60 minutes before ESWL, followed by 400 mg every 8 hours for the first 24 hours after the procedure (total of three doses), in accordance with standard clinical practice. Participants will be allowed to receive rescue analgesia according to the study protocol if pain is not adequately controlled.
  Arms: Ibuprofen Group

SUMMARY:
Pain after extracorporeal shock wave lithotripsy (ESWL), a non-surgical procedure used to treat kidney stones, is common and is usually treated with non-steroidal anti-inflammatory drugs (NSAIDs) such as ibuprofen. However, NSAIDs may cause side effects in some patients, including stomach irritation and kidney problems.

Palmitoylethanolamide (PEA) is a naturally occurring substance in the body with anti-inflammatory and pain-relieving properties and has been shown to be safe in previous studies. This study aims to compare the effectiveness of PEA with ibuprofen for controlling acute postoperative pain after ESWL.

Participants undergoing ESWL will be randomly assigned to receive either oral PEA or oral ibuprofen. Pain intensity will be measured using a visual analogue scale during the first 24 hours after the procedure. The use of rescue pain medication and any side effects will also be recorded.

The results of this study may help determine whether PEA can be an effective alternative to ibuprofen for the management of acute pain after ESWL.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* ASA I or II
* Undergoing elective ESWL for renal or upper ureteric calculi
* Expected discharge same day or within 24 hours (outpatient ESWL).
* Able to provide informed consent and comply with study procedures (including diary/VAS recordings).
* Not currently taking chronic NSAIDs, opioids, or PEA supplements for ≥7 days prior to ESWL.

Exclusion Criteria:

* Chronic pain or daily analgesic use.
* Known allergy or contraindication to PEA, ibuprofen.
* Active peptic ulcer disease, known bleeding disorder, anticoagulant therapy
* Pregnancy or lactation.
* Use of steroids or other pain-modulating drugs.
* Severe renal impairment (eGFR <30 mL/min/1.73 m²).
* Hepatic failure or significant liver enzyme elevation (AST/ALT >3× ULN).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity measured by Visual Analogue Scale (VAS) | 2 hours after ESWL
  Pain intensity will be assessed using a 10-cm visual analogue scale (VAS), where 0 indicates no pain and 10 indicates the worst imaginable pain. The primary comparison will be the VAS score measured 2 hours after extracorporeal shock wave lithotripsy (ESWL) between the palmitoylethanolamide and ibuprofen groups.

SECONDARY OUTCOMES:
Pain intensity over the first 24 hours after ESWL | From recovery room arrival up to 24 hours after ESWL
  Pain intensity will be assessed using the 10-cm visual analogue scale (VAS) at predefined time points after ESWL (e.g., recovery room, 30 minutes, 1 hour, 4 hours, 6 hours, 12 hours, and 24 hours) to evaluate pain progression over time.
Time to first rescue analgesia | Up to 24 hours after ESWL
  Time elapsed (in minutes) from completion of ESWL to the first administration of rescue analgesic medication for uncontrolled pain.
Total rescue analgesic consumption within 24 hours | Up to 24 hours after ESWL
  Total amount of rescue analgesics administered within the first 24 hours after ESWL, recorded as grams of paracetamol and opioid consumption converted to morphine milligram equivalents (MME), if applicable.
Proportion of patients achieving clinically meaningful pain relief | Within 24 hours after ESWL
  The proportion of participants achieving at least a 30% and 50% reduction in pain intensity on the VAS compared with baseline or peak postoperative pain.
Incidence of adverse events | From first dose of study medication up to 7 days after ESWL
  The number and type of adverse events related to study medications, including gastrointestinal symptoms, renal-related symptoms, allergic reactions, or any other reported side effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University Hospital, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided